CLINICAL TRIAL: NCT04019314
Title: Assessment of ProEnkephalin to Detect Acute Kidney Injury (AKI) in Patients Hospitalized for Volume Overload Decompensated Chronic Heart Failure
Brief Title: Assessment of ProEnkephalin to Detect Acute Kidney Injury (AKI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Sphingotec GmbH (Industry)
Responsible Party: Principal Investigator, Wayne L. Miller, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 18-000181
Record Dates: First submitted 2019-06-25; First posted 2019-07-15 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure; Volume Overload; Decompensated Heart Failure; Systolic Heart Failure
MeSH Terms: conditions — Heart Failure; Edema; Heart Failure, Systolic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with know chronic systolic heart failure (Experimental): Subjects with know chronic systolic heart failure (LVEF<50%) admitted to SMH Heart Failure Medical Service for decompensated HF with clinical findings of volume overload requiring advanced diuretic therapy intervention and management will receive daily blood draws and quantitative blood volume analysis
  Interventions: Procedure: Blood Collection; Procedure: Blood Volume Analysis

INTERVENTIONS:
Procedure: Blood Collection — Samples for proEnkephalin PENK will be obtained daily and aliquots of these samples will be stored for later batch assays.
Procedure: Blood Volume Analysis — A small amount of a radioactive isotope or tracer is injected and blood samples are taken at 6 time points during the test and analyzed.

SUMMARY:
Researchers are observing the values of proEnkephalin (PENK) via a blood draw in hospitalized patients that are volume overloaded requiring diuresis. If changes in PENK are found, physicians may predict values of change in kidney function during treatment.

DETAILED DESCRIPTION:
The purpose of this study will be to probe if values of proEnkephalin, called PENK in this proposal, can identify those patients who develop AKI. This biomarker is an opioid that is rapidly released in response to renal injury. At a cut-off value of 100pmol/L, it has been reported to have excellent sensitivity and specificity for detecting renal injury. PENK has been shown to be prognostic of WRF and outcomes in patients with acute heart failure but requires evaluation of efficacy in detecting AKI in standard of care clinical practice settings. In this study we propose to evaluate the baseline presence of plasma and/or serum levels of biomarkers of renal injury and changes in these biomarkers during the course of in-hospital intravenous diuretic therapy. The question is if threshold values of the biomarkers can be identified and if those threshold values would indicate a clinically significant change in renal function that would warrant a change in diuretic therapy to occur. In this context the quantitative assessment of intravascular volume will provide objective corroboration as to volume status in relation to biomarker levels and changes during treatment. If this approach can be proven to be fruitful, it would be anticipated that a subsequent study, a clinical trial, to test the hypothesis that biomarkers of AKI, specifically PENK, could be used to identify and avoid AKI in hospitalized patients with decompensated HF.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* LVEF <50% measured within 6 months of index hospitalization
* Clinically identified volume overload with at least one sign of volume overload (pre-admission fluid weight gain, edema, increased DOE, PND, orthopnea, JVD on examination) and a need for intravenous diuretic therapy

Exclusion Criteria:

* Baseline sCr >3.0mg/dL and K+ <3.0 and >5.5mEq/L
* Hemoglobin < 9.0g/dL
* Systemic systolic blood pressure consistently <100mm Hg
* Patients being treated with hemodialysis, CKD stage 5 or s/p renal transplantation
* S/P cardiac transplant or LVAD implantation/total artificial heart
* Pregnancy or of child bearing potential
* Allergy to iodine
* Unable to provide informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Assessment of ProEnkephalin to detect acute kidney injury in hospitalized to identify baseline values of PENK biomarkers of AKI in relation to measured intravascular volume. | Hospital admission through hospital discharge, approximately 6 days
  Blood samples obtained during admission will be assessed for PENK biomarkers. Samples will be stored from all subjects for future analysis if PENK is supportive of a trend based on the PENK data.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Miller, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials